CLINICAL TRIAL: NCT05626153
Title: Effects of Anesthesia Quality Improvement on Outcomes of Patients With Planned ICU Admission: a Prospective Pre-post Intervention Study
Brief Title: Anesthesia Quality Improvement and Patients With Planned ICU Admission
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2022-413
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia; Extubation; Intensive Care Unit; Postoperative Complications
Keywords: Anesthesia management; Early extubation; Intensive care unit admission; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine anesthesia care (Active Comparator): • Implementing anesthesia management according to current routine practice.
  Interventions: Other: Routine anesthesia care
- Improved anesthesia care (Experimental): * Encourage regional anesthesia or combined regional-general anesthesia.
  * Encourage goal-directed fluid therapy, lung-protective ventilation, and active warming during surgery.
  * Encourage extubation in the operating room at the end of surgery.
  * Encourage multimodal analgesia after surgery.
  * Encourage strict indication for ICU admission after surgery.
  Interventions: Other: Improved anesthesia care

INTERVENTIONS:
Other: Routine anesthesia care — • Implementing anesthesia management according to current routine practice.
  Arms: Routine anesthesia care
Other: Improved anesthesia care — * Encourage regional anesthesia or combined regional-general anesthesia.
  * Encourage goal-directed fluid therapy, lung-protective ventilation, and active warming during surgery.
  * Encourage extubation in the operating room at the end of surgery.
  * Encourage multimodal analgesia after surgery.
  * Encourage strict indication for ICU admission after surgery.
  Arms: Improved anesthesia care

SUMMARY:
Intensive care unit (ICU) is an important part of perioperative management for high-risk patients but is associated with higher medical costs. Improper ICU admission may produce overtreatment without beneficial effects. In clinical practice, delayed recovery after general anesthesia is a common indication for ICU admission after surgery. The concept of Enhanced Recovery After Surgery recommends early extubation. The investigators suppose that, for patients with planned ICU admission after elective surgery, implementing anesthesia quality improvement including extubation in the operating room will reduce the rate of ICU admission after surgery without increasing complications.

DETAILED DESCRIPTION:
Intensive care unit (ICU) is an important part of perioperative management for high-risk patients but is associated with higher medical costs. Improper ICU admission may produce overtreatment without beneficial effects. Studies found that immediate ICU admission after surgery did not reduce the perioperative mortality. Some authors suggested that the indication of ICU admission should be the occurrence of postoperative complications, which will reasonably reduce the use of medical resources.

In clinical practice, delayed recovery after general anesthesia is a common indication for ICU admission after surgery. Old age, high ASA grade, respiratory complications, long duration surgery, large-volume fluid infusion, and use of vasopressors were main factors associated with delayed recovery. The concept of Enhanced Recovery After Surgery recommends early extubation after surgery. Studies showed that, for patients after organ transplantation, immediate extubation in the operating room can shorten hospital stay and reduce medical costs, without increasing mortality.

The investigators suppose that, for patients with planned ICU admission after elective surgery, implementing anesthesia quality improvement including extubation in the operating room will reduce the rate of ICU admission after surgery without increasing postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Scheduled to undergo elective surgery.
* Planned ICU admission after surgery.

Exclusion Criteria:

* Refused to participate in the study.
* ICU admission before surgery.
* Unexpected ICU admission.
* Other conditions that are considered unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative complication | Up to 30 days after surgery
  Postoperative complications are defined as newly occurred medical conditions that are considered harmful to patients' recovery and require therapeutic intervention, that is grade II or higher on Clavin-Dindo classification.

SECONDARY OUTCOMES:
Rate of ICU admission | On the 1 day of surgery
  Rate of ICU admission
Incidence of postoperative delirium | Up to 5 days after surgery
  Delirium is assessed with the Three-dimensional Confusion Assessment Method (3D-CAM) twice daily (8:00-10:00 am and 18:00-20:00 pm).
Rate of delayed neurocognitive recovery | up to 7 days after surgery
  Cognitive function is assessed with the Montreal Cognitive Assessment (MoCA) before surgery and at discharge. A decrease of 1 standard deviation (SD) or more from baseline is defined as the development of delayed neurocognitive recovery.
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Medical costs during hospitalization | Up to 30 days after surgery
  Medical costs during hospitalization

OTHER OUTCOMES:
Duration of mechanical ventilation | up to 30 days after surgery
  Duration of mechanical ventilation
Length of stay in ICU after surgery | Up to 30 days after surgery
  Length of stay in ICU after surgery
Rate of ICU re-admission | Up to 30 days after surgery
  ICU re-admission is defined as ICU admission from the general wards after surgery
All-cause 30-day mortality | Up to 30 days after surgery
  All-cause 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahan BC, Koulenti D, Arvaniti K, Beavis V, Campbell D, Chan M, Moreno R, Pearse RM; International Surgical Outcomes Study (ISOS) group. Critical care admission following elective surgery was not associated with survival benefit: prospective analysis of data from 27 countries. Intensive Care Med. 2017 Jul;43(7):971-979. doi: 10.1007/s00134-016-4633-8. Epub 2017 Apr 25. PMID 28439646
- [Background] Vourc'h M, Asehnoune K. Postoperative admission in surgical ICU, less is more? Anaesth Crit Care Pain Med. 2019 Jun;38(3):217-219. doi: 10.1016/j.accpm.2019.03.006. Epub 2019 Apr 2. No abstract available. PMID 30951884
- [Background] Zampieri FG. Elective ICU admission after major surgery: can too much support be futile? J Thorac Dis. 2018 Jun;10(Suppl 17):S1992-S1994. doi: 10.21037/jtd.2018.05.154. No abstract available. PMID 30023100
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Anastasian ZH, Gaudet JG, Levitt LC, Mergeche JL, Heyer EJ, Berman MF. Factors that correlate with the decision to delay extubation after multilevel prone spine surgery. J Neurosurg Anesthesiol. 2014 Apr;26(2):167-71. doi: 10.1097/ANA.0000000000000028. PMID 24296539
- [Background] Li F, Gorji R, Tallarico R, Dodds C, Modes K, Mangat S, Yang ZJ. Risk factors for delayed extubation in thoracic and lumbar spine surgery: a retrospective analysis of 135 patients. J Anesth. 2014 Apr;28(2):161-6. doi: 10.1007/s00540-013-1689-2. Epub 2013 Aug 9. PMID 23934263
- [Background] David RA, Brooke BS, Hanson KT, Goodney PP, Genovese EA, Baril DT, Gloviczki P, DeMartino RR. Early extubation is associated with reduced length of stay and improved outcomes after elective aortic surgery in the Vascular Quality Initiative. J Vasc Surg. 2017 Jul;66(1):79-94.e14. doi: 10.1016/j.jvs.2016.12.122. Epub 2017 Mar 31. PMID 28366307
- [Background] Gal J, Hunter S, Reich D, Franz E, DeMaria S, Neifert S, Lin HM, Liu X, Caridi J, Katz D. Delayed extubation in spine surgery is associated with increased postoperative complications and hospital episode-based resource utilization. J Clin Anesth. 2022 May;77:110636. doi: 10.1016/j.jclinane.2021.110636. Epub 2021 Dec 20. PMID 34933241
- [Background] Stumpo V, Staartjes VE, Quddusi A, Corniola MV, Tessitore E, Schroder ML, Anderer EG, Stienen MN, Serra C, Regli L. Enhanced Recovery After Surgery strategies for elective craniotomy: a systematic review. J Neurosurg. 2021 May 7;135(6):1857-1881. doi: 10.3171/2020.10.JNS203160. Print 2021 Dec 1. PMID 33962374
- [Background] Brustia R, Monsel A, Skurzak S, Schiffer E, Carrier FM, Patrono D, Kaba A, Detry O, Malbouisson L, Andraus W, Vandenbroucke-Menu F, Biancofiore G, Kaido T, Compagnon P, Uemoto S, Rodriguez Laiz G, De Boer M, Orloff S, Melgar P, Buis C, Zeillemaker-Hoekstra M, Usher H, Reyntjens K, Baird E, Demartines N, Wigmore S, Scatton O. Guidelines for Perioperative Care for Liver Transplantation: Enhanced Recovery After Surgery (ERAS) Recommendations. Transplantation. 2022 Mar 1;106(3):552-561. doi: 10.1097/TP.0000000000003808. PMID 33966024
- [Background] Feltracco P, Serra E, Barbieri S, Milevoj M, Salvaterra F, Marulli G, Ori C. Noninvasive ventilation in adult liver transplantation. Transplant Proc. 2008 Jul-Aug;40(6):1979-82. doi: 10.1016/j.transproceed.2008.05.006. PMID 18675106
- [Background] Xu Y, Zuo Y, Zhou L, Hao X, Xiao X, Ye M, Bo L, Jiang C, Yang J. Extubation in the operating room results in fewer composite mechanical ventilation-related adverse outcomes in patients after liver transplantation: a retrospective cohort study. BMC Anesthesiol. 2021 Nov 18;21(1):286. doi: 10.1186/s12871-021-01508-1. PMID 34794387
- [Background] Khwannimit B, Bhurayanontachai R. Prediction of fluid responsiveness in septic shock patients: comparing stroke volume variation by FloTrac/Vigileo and automated pulse pressure variation. Eur J Anaesthesiol. 2012 Feb;29(2):64-9. doi: 10.1097/EJA.0b013e32834b7d82. PMID 21946822
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912